CLINICAL TRIAL: NCT01935245
Title: Platelet Function in Minimal Extracorporeal Circulation Versus Conventional Extracorporeal Circulation in Coronary Artery Bypass Grafting
Brief Title: Platelet Function in Minimal Extracorporeal Circulation in CABG
Acronym: ECCTEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Ingeborg Herold, MD, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL40546.060.12
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Thrombocytopathy
Keywords: Coronary artery bypass grafting; Extracorporeal circulation; Minimal extracorporeal circulation; Coagulopathy; Thrombocytopathy; Platelet dysfunction
MeSH Terms: conditions — Blood Platelet Disorders; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mini extracorporeal circulation (Experimental): Patients undergoing coronary artery bypass surgery on minimal extracorporeal circulation
  Interventions: Device: Mini extracorporeal circulation
- Conventional extracorporeal circulation (Active Comparator): Patients undergoing coronary artery bypass surgery on conventional extracorporeal circulation
  Interventions: Device: Conventional extracorporeal circulation

INTERVENTIONS:
Device: Mini extracorporeal circulation — Minimal-ECC versus conventional ECC circuits minimise foreign surface-blood interaction and are heparinized from tip to tip. The tubing length has been shortened to decrease crystalloid prime. Cardiotomy suction is minimised, which leads to less fibrinolysis. An active air-removal device is added to the closed circuit.
  The use of minimal ECC has already shown a significant reduction of the systemic inflammatory reaction and less peroperative transfusion of blood products.
  Other Names: Mini- ECC: ECC.O Oxygenator
  Arms: Mini extracorporeal circulation
Device: Conventional extracorporeal circulation
  Other Names: Conventional ECC: D903 Avant Oxygenator
  Arms: Conventional extracorporeal circulation

SUMMARY:
Rationale:

Cardiac surgery with extracorporeal circulation (ECC) triggers platelets. Minimal extracorporeal circulation system (minimal-ECC) has several advantages compared with conventional ECC amongst less platelet activation. Platelet function can be analysed with thromboelastography (TEG) and multiple electrode aggregometry (MEA).

Objective:

The use of minimal ECC leads to less platelet dysfunction compared with conventional ECC in coronary artery bypass grafting (CABG) analysed with TEG and MEA

Study design:

Single center, prospective, randomized, pilot study

Study population:

Group 1:

20 patients undergoing CABG using minimal ECC. Patients continued the use of acetylsalicylic acid and discontinued the use of clopidogrel minimal 5 days preoperative.

Group 2:

20 patients undergoing CABG using conventional ECC. Patients continued the use of acetylsalicylic acid and discontinued the use of clopidogrel minimal 5 days preoperative.

Intervention:

Group 1: CABG using minimal ECC Group 2: CABG using conventional ECC

Main study parameters/endpoints:

1. Results of TEG and MEA, see detailed description
2. Per operative blood loss and total blood loss 24 hours after CABG
3. Total amount of transfused platelet units during CABG and 24 hours after CABG

DETAILED DESCRIPTION:
Platelet function test

Thromboelastography (TEG) TEG is a test which provides information on the complete haemostasis. Also fibrinolysis can be measured. The strength of the clot can be measured. This provides information about platelet concentration, -function and platelet-fibrin interaction. It is measured in a medium with added heparinase, an enzyme that degrades heparin,, which makes TEG measurement possible during ECC. The results from the TEG will be displayed graphically and numerically. The letter R (reaction time) represents the time before the clot formation starts. This time is predominately dependent on coagulation factors and inhibitors such as heparin. The velocity at which the clot is then formed is displayed as the letter K (time between 2 mm en 20 mm amplitude in the thromboelastogram). The firmness of the clot is the maximum amplitude in the thromboelastogram (MA) and is dependent on the amount and function of the thrombocytes, fibrinogen concentration and factor XIII concentration of the sample. Fibrinolysis will be visualised in the parameter that displays the velocity of dissolving the clot (LY30= fibrinolysis 30 minutes after MA).

In case of a severe coagulation factor independency or use of heparin, the R parameter will be elongated. In severe thrombocytopathy, thrombocytopenia or a low fibrinogen concentration the graphic will show a lowered MA. In hyperfibrinolysis the LY30 will be elongated.

Multiple electrode Aggregometry (MEA) MEA is a technique to test platelet function in whole blood based on classical impedance aggregometry. The use of whole blood makes centrifugation redundant. The use of agonist ADP, arachidonic acid, collagen and TRAP provides information about platelet aggregation, and simultaneously provides specific information of the routes inhibited by clopidogrel and acetylsalicylic acid.

MEA calculates three parameters. The most important parameter, the area under the curve (AUC), reflexes the overall platelet activity . The area under the curve is influenced by the total height of the aggregation curve as well as by its slope. The other parameters are the height of the curve that describes the aggregation. The maximum slope of the curve describes the reflex velocity.

Results TEG and MEA contain:

* TEG angle
* TEG K
* TEG LY 30
* TEG MA
* TEG R

MEA:

* MEA adenosine diphosphate (ADP)
* MEA arachidonic acid
* MEA collagen
* MEA thrombin receptor activating peptide (TRAP)

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass grafting
* Use of acetylsalicylic acid
* > 18 years
* body surface area < 2.1 [M2]

Exclusion Criteria:

* Emergency procedures
* Platelet function disorders
* Clopidogrel stopped < 5 days
* Thrombocytes < 150/ nanoliter
* Renal insufficiency, creatinin clearance <60 ml/min
* Chronic alcohol abuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Platelet function | Post-cardiopulmonary bypass
  Change in thrombocyte function is measured directly after Protamine and three hours after operation. This change is correlated to the reference preoperatively.

SECONDARY OUTCOMES:
Perioperative blood loss | 24 hours

OTHER OUTCOMES:
Amount of platelet or fresh frozen plasma transfusion | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg HF Herold, MD, Principal Investigator — Catharina hospital Eindhoven, The Netherlands
Locations (1):
- Catharina hospital Eindhoven, Eindhoven, North Brabant, Netherlands